CLINICAL TRIAL: NCT01063738
Title: Rehabilitating Muscle After Intensive Care
Acronym: REMAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Helens & Knowsley Teaching Hospitals NHS Trust (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB_PG_1208_18030
Record Dates: First submitted 2010-02-02; First posted 2010-02-05 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Recovery From Critical Illness
Keywords: Rehabilitation; Intensive Care; Critical illness; Physiotherapy; Nutritional supplementation
MeSH Terms: conditions — Critical Illness | interventions — Intensive Care Units

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ICU Recovery Manual & placebo supplement (Active Comparator): Patients will receive the standard self-directed rehabilitation package and a placebo nutritional supplement
  Interventions: Other: Intensive Care Unit (ICU) Recovery Manual; Dietary Supplement: Placebo nutritional supplement
- ICU recovery manual & amino acid (AA) supplement (Experimental): Patients will receive the standard self-directed rehabilitation package with the essential amino acid supplement
  Interventions: Dietary Supplement: Amino acid supplement; Other: Intensive Care Unit (ICU) Recovery Manual
- PEPSE & placebo supplement (Experimental): Patients will receive the standard self-directed rehabilitation package plus PEPSE and the placebo nutritional supplement
  Interventions: Other: PEPSE; Other: Intensive Care Unit (ICU) Recovery Manual; Dietary Supplement: Placebo nutritional supplement
- PEPSE & AA supplement (Experimental): Patients will receive the standard self-directed rehabilitation package plus PEPSE and the essential amino acid nutritional supplement
  Interventions: Dietary Supplement: Amino acid supplement; Other: PEPSE; Other: Intensive Care Unit (ICU) Recovery Manual

INTERVENTIONS:
Dietary Supplement: Amino acid supplement — Flavoured essential amino acid supplement and glutamine dipeptide taken twice daily for 3 months
  Arms: ICU recovery manual & amino acid (AA) supplement; PEPSE & AA supplement
Other: PEPSE — Enhanced physiotherapy programme of 3 1 hour sessions per week for 6 weeks while in hospital and once discharged home 1 supervised outpatient session of 1 hour and 2 home exercise sessions per week (PEPSE).
  Arms: PEPSE & AA supplement; PEPSE & placebo supplement
Other: Intensive Care Unit (ICU) Recovery Manual — Standard self-directed 6 week rehabilitation package
Dietary Supplement: Placebo nutritional supplement — Cherry flavoured low calorie and low protein placebo drink
  Arms: ICU Recovery Manual & placebo supplement; PEPSE & placebo supplement

SUMMARY:
The study will examine the effect of amino acid supplements and enhanced physiotherapy on physical recovery following critical illness in intensive care.

DETAILED DESCRIPTION:
Critically ill patients aged 45 years and over will be recruited during recovery after intensive care. Using a randomised controlled, blind at follow-up design the study will examine whether the combination of an amino acid supplement and an enhanced physiotherapy programme improve the rehabilitation of muscle following intensive care better than a self-guided rehabilitation programme alone or with either an amino acid supplement or the enhanced physiotherapy programme. The Primary efficacy outcome will be the improvement in six minute walking test measured at 3 months post intensive care discharge. Secondary efficacy parameters will be insulin resistance, health related quality of life and muscle mass using DEXA scanning at 3 months and 1 year post intensive care discharge.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age and over with an intensive care stay of five days or more

Exclusion Criteria:

* Physically not capable of engaging with the practical requirements of the study

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-08; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The change in the distance walked by patients in 6 minutes (6 minute walk test) between recruitment to the study and 3 months post intensive care discharge | 3 months

SECONDARY OUTCOMES:
Improvement in insulin resistance between recruitment to the study and the 1 year follow-up point | 1 year
Improvement in patients perception of their health related quality of life between recruitment to the study and the 1 year follow-up point | 1 year
Increase in muscle mass and bone density assessed using dual energy x-ray absorptiometry (DEXA) scanning between recruitment to the study and the 1 year follow-up point | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Griffiths, MD, Principal Investigator — St Helens & Knowley Teaching NHS Trust
Locations (2):
- United Kingdom (2):
  - St Helens & Knowsley Teaching NHS Trust, Prescot, Merseyside
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Jones C, Eddleston J, McCairn A, Dowling S, McWilliams D, Coughlan E, Griffiths RD. Improving rehabilitation after critical illness through outpatient physiotherapy classes and essential amino acid supplement: A randomized controlled trial. J Crit Care. 2015 Oct;30(5):901-7. doi: 10.1016/j.jcrc.2015.05.002. Epub 2015 May 9. PMID 26004031